CLINICAL TRIAL: NCT00400140
Title: Pilot Study to Assess the Efficacy of Short Exposure to Defocus to Slow the Progression of Myopia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other)
Responsible Party: Audrey Chia, Singapore National Eye Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R473/22/2006
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia
Keywords: Myopia, defocus
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- A (Experimental)
  Interventions: Device: Hyperopic lens

INTERVENTIONS:
Device: Hyperopic lens — +3 D glasses

SUMMARY:
The objective of this pilot study is to establish whether brief periods of high levels of acutely imposed myopic defocus can be used to slow the progression of myopia in children, as measured by changes in spherical equivalent refraction and axial length.

DETAILED DESCRIPTION:
Recent results on animal models of myopia suggest that the eye has the ability to detect the overall sign of defocus of images falling on the retina, with myopic defocus imposed by the fitting of plus-lenses halting or slowing axial elongation of the eye. In the animal models, these STOP growth signals have been shown to be particularly strong - with brief periods of high myopic defocus able to outweigh the effects of prolonged periods of imposed hyperopic defocus in promoting eye growth. These results therefore suggest a novel strategy for preventing the progression of myopia in children - the imposition of high levels of myopia for brief periods of time. This approach is conceptually distinct from under-correction, which imposes chronic mild myopic defocus.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 to 12 years
2. Refractive error of spherical equivalent -1.00 D to -6.00D in each eye as measured by cycloplegic autorefraction
3. Active myopia progression of at least spherical equivalent -0.50 D over the last 12 months as determined or suggested by refractive records or change in lens power
4. Astigmatism of less than or equal to -1.50 D as measured by non-cycloplegic or cycloplegic autorefraction
5. Distance vision correctable to logMAR 0.1 or better in both eyes
6. Normal intraocular pressure of not greater than 21 mmHg
7. Normal ocular health other than myopia
8. In good general health
9. Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

1. Baseline Anisometropia of > 1.5D
2. Ocular or systemic diseases which may affect vision or refractive error
3. Defective binocular function or stereopsis
4. Amblyopia or manifest strabismus including intermittent tropia
5. Previous or current use of atropine or pirenzepine
6. Any other conditions precluding adherence to the protocol including unwillingness to refrain from contact lens wear for the duration of the study
7. Allergy to cyclopentolate, proparacaine and benzalkonium chloride

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Myopia progression as measured by spherical equivalent, and axial length | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Chia, FRANZCO, Principal Investigator — Singapore National Eye Center
Locations (1):
- SNEC, Singapore, Singapore